CLINICAL TRIAL: NCT04391985
Title: Retreatment Efficacy of Sofosbuvir/Ombitasvir/Paritaprevir/ Ritonavir + Ribavirin for Hepatitis C Virus Genotype 4 Patients
Brief Title: Sofosbuvir/Ombitasvir/Paritaprevir/ Ritonavir and Ribavirin for Hepatitis C Virus Genotype 4 Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Abdel-Gabbar, Ph.D, Associate Prof, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Qu-RBV
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Chronic Hepatitis C Virus Infection
Keywords: Sofosbuvir; Ombitasvir; Paritaprevir; Ribavirin; Ritonavir; HCV GT 4; Experienced Egyptian Patients; Cirrhotic; Non-Cirrhotic
MeSH Terms: interventions — paritaprevir; ombitasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cirrhotic Participants (Active Comparator): The experienced participants(113 participants) who failed prior DAA treatments. They were allocated to cirrhotic (30 participants) and treated for 12 weeks.
  Interventions: Drug: SOF plus (OBV/PTV/r) plus RBV
- Non-cirrhotic Participants (Active Comparator): The experienced non-cirrhotic participants(83 participants) who failed prior DAA treatments. They were treated for 12 weeks.
  Interventions: Drug: SOF plus (OBV/PTV/r) plus RBV

INTERVENTIONS:
Drug: SOF plus (OBV/PTV/r) plus RBV — They were given SOF in a dose of 400 mg/day, and a fixed dose combination of OBV (25 mg), PTV (150 mg), and r (100 mg) taken with food once daily. RBV was supplied in 200 mg capsules, and the recommended dose was 600 mg/ day to reach 1200 mg/day based on patient's body weight and tolerability.
  Other Names: Paritaprevir (ABT-450) is inhibitor of the NS3-4A serine protease; Sovaldi is a trade name of sofosbuvir; Ombitasvir (ABT 267) is an NS5A inhibitor

SUMMARY:
enrolled participants were treated orally with SOF plus a fixed dose combination of OBV/PTV/r plus RBV.

DETAILED DESCRIPTION:
Enrolled participants were treated orally with SOF plus a fixed dose combination of Sofosbuvir/Ombitasvir/Paritaprevir/ Ritonavir plus Ribavirin (OBV/PTV/r plus RBV), which was administered orally based on the participants' tolerability. The primary end point was a sustained virological response (HCV RNA level < 15 IU/ mL), observed 12 weeks after the end of the treatment (SVR12).

ELIGIBILITY:
Inclusion Criteria:

* The experienced participants who were treated previously with (SOF/DCV) , (SOF/SMV), (SOF/RBV), or (SOF/pegINF/RBV).
* The presence of compensated liver cirrhosis was documented by ultrasonographic examination, liver biopsy, results of Fibroscan or FIB-4 score, and laboratory markers, like FIB-4 > 3.25 (advanced fibrosis or cirrhosis), albumin < 3.5, total bilirubin > 1.2, and also confirmed by clinical characteristics such as lower limb edema, splenomegaly, esophageal varices.

Exclusion Criteria:

* liver disease of non-HCV GT4 etiology, coinfection with hepatitis B or HIV
* poorly controlled diabetes (HbA1C > 8)
* participants, hepatocellular carcinoma, a history of extrahepatic malignancy in the 5 years prior to the study
* renal failure
* evidence of hepatic decompensation
* blood picture abnormalities such as anemia (hemoglobin concentration of < 10 g/dL)
* thrombocytopenia (platelets count < 50,000 cells/mm3).
* major severe illness such as congestive heart failure and respiratory failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) in Each Treatment Arm | 12 weeks after last dose
  SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) level < 15 IU/ml 12 weeks after the last dose of drugs.
Number of Participants With Adverse Events in Each Treatment Arm | Screening up to 12 weeks after last dose]
  An adverse event (AE) is defined as any untoward medical occurrence in a participant clinical investigation after administering a pharmaceutical drugs Serious adverse event (SAE) is an event that results in death, life-threatening, requires hospitalization, or significant disability/incapacity

SECONDARY OUTCOMES:
Percentage of Participants With Viral relapse | Up to 12 weeks after last dose
  Viral relapse was HCV RNA level undetectable at End of Treatment (EOT) (≤ 15 IU/ml), but detectable HCV RNA ( > 15 IU/ml) levels 12 weeks after planned EOT.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdel-Moneim A, Aboud A, Abdel-Gabbar M, Zanaty M, Ramadan M. Retreatment Efficacy of Sofosbuvir/Ombitasvir/Paritaprevir/Ritonavir + Ribavirin for Hepatitis C Virus Genotype 4 Patients. Dig Dis Sci. 2018 May;63(5):1341-1347. doi: 10.1007/s10620-018-5005-8. Epub 2018 Mar 15. PMID 29546644
- See also: This link clarify the retreatment efficacy and safety of the SOF with OBV/PTV/r + RBV, for chronic HCV GT4-experienced patients who failed treatment with DAA-based regimens. — https://link.springer.com/article/10.1007/s10620-018-5005-8